CLINICAL TRIAL: NCT03111329
Title: A Prospective, Randomized and Controlled Trial Comparing the Role of no Gastric Residual ASSessment and Standard Gastric Residual Measurement for the Achievement of Full Enteral Feeding in Preterm Infants
Brief Title: Does Routine Assessment of Gastric Residuals in Preterm Neonates Influence Time Taken to Reach Full Enteral Feeding?
Acronym: GRASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Collaborators: Coombe Women and Infants University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GRASS-1
Record Dates: First submitted 2017-03-23; First posted 2017-04-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Gastric Residuals Assessment; Prematurity; Sepsis Newborn; Necrotizing Enterocolitis of Newborn
Keywords: Gastric residuals assessment; Prematurity; Necrotizing Enterocolitis of Newborn; Sepsis Newborn; Nutrition of newborn; feeding tolerance of newborn
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Randomization into 2 groups (interventional and control) with crossover rescue strategy.
Who Masked: Outcomes Assessor
Masking Description: Open label during intervention, assessor of outcomes will be blinded to group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRASS - Intervention group (Experimental): The intervention group (GRASS) will receive 3 hourly feeds, with no gastric residuals being aspirated. Solely opening of the nasogastric tube once every 6 hours to relieve possible backflow of gastric content will be allowed. Amount of enteral feeds given and increase in dose will be specified in an enteral feeding plan prior to start of the study. Amount of enteral feeds given will increase every six hours with a calculated overall increase of 20 ml/kg of birth weight in the total amount given every 24 hours.
  Intervention = NO aspiration of gastric residuals
  Interventions: Other: No aspiration of gastric residuals
- Standard Approach group (No Intervention): Standard Approach group serving as control group will be treated as per standard approach - participants will be fed 3 hourly and gastric residuals checked via nasogastric tube prior to each feed. Amount of enteral feeds given and increase in dose will be specified in an enteral feeding plan prior to start of the study. Amount of enteral feeds given will increase every six hours with a calculated overall increase of 20 ml/kg of birth weight in the total amount given every 24 hours.

INTERVENTIONS:
Other: No aspiration of gastric residuals — No assessment of gastric residuals will be performed prior to administering 3-hourly feeds with increasing amounts of the feeds given as per a predefined plan
  Arms: GRASS - Intervention group

SUMMARY:
The study aims to compare routine assessment of gastric residuals versus no assessment of residuals in preterm neonates with respect to time taken for achieving full enteral feeding and the incidence of possible complications, such as feeding intolerance, necrotizing enterocolitis, sepsis etc.

DETAILED DESCRIPTION:
In general, regular assessment of gastric residuals and its´ evaluation prior to every feeding is considered standard practice for preterm neonates in neonatal intensive care units. It is believed useful to confirm correct placement of the orogastric or nasogastric tube and thought of as necessary to aid the decision of enteral feeding advancement by informing about possible remains of contents from previous feeding. Furthermore, evaluation of gastric residuals is routinely performed in order to assess for feeding intolerance and used as a possible indicator of risk for development of necrotizing enterocolitis.

However there is conflicting evidence to support the approach of routine gastric residuals assessment and it seems unclear whether it confers any clinical benefit. Withholding of enteral feeding or cessation of advancement in the amounts given due to misinterpretation of routine gastric aspirates may have a negative impact on the preterm neonate. This can potentially involve prolonged indwelling of venous catheters, higher risk of infection and growth restriction with potentially worse developmental outcome in particular for very low birth weight infants.

This randomized controlled clinical study aims to compare a control group with regular assessment and evaluation of gastric residuals and an intervention group with no routine assessment of residuals prior to feeding advancement, for the time taken to reach full enteral feeding and for occurrence of any observed complications including necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate, born between 26+0 and 30+0 weeks of gestation
* Birth weight below 1500g
* Parental informed consent obtained

Exclusion Criteria:

* Intrauterine growth retardation (birth weight below 5th centile for given gestational age and gender)
* Life-threatening events requiring full resuscitation at the delivery room (severe hypoxia, bleeding), and persistently raised lactate value of more than 5 mmol/l
* Circulatory instability requiring treatment with inotropes
* Highly suspected early onset sepsis with alteration of general clinical state, in particular with worsened peripheral perfusion and circulatory decompensation prior to study begin (during the first 6 hours after admission to NICU)
* Known malformations of gastrointestinal tract, known diagnosis of congenital diaphragmatic hernia, any other life-limiting serious congenital malformations

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Number of days taken to achieve full enteral feeding (i.e. dose of 100ml/kg/day) | 5 days after delivery for yes or no answer to whether full enteral feeding has been achieved, thereafter daily for the first three weeks until full enteral feeding has been reached
  Time taken (in hours) to reach full enteral feeding, defined as overall dose of 100ml of feeds/kg of birth weight/ day

SECONDARY OUTCOMES:
Withholding of enteral feeding | Through first (on average) two to three weeks of the study until full enteral feeding is achieved.
  The need to withhold enteral feeds due to clinical situation as per clinical judgement of the clinician in charge
Total duration of parenteral infusion | Through first (on average) two to three weeks of the study until full enteral feeding is achieved.
  The length of time (in hours) that parenteral infusion is needed
Total duration of indwelling central venous catheter | Through first (on average) two to three weeks of the study until full enteral feeding is achieved.
  The length of time (in hours) that an indwelling central venous catheter is needed
Hypoglycaemia | Through first (on average) two to three weeks of the study until full enteral feeding is achieved.
  Any episodes of hypoglycaemia (value less than 2,5 mmol/l) after attainment of full enteral feeding
Late onset sepsis | Duration of hospitalization, an average of 8-15 weeks
  The incidence of late onset sepsis
Necrotizing enterocolitis | Duration of hospitalization, an average of 8-15 weeks
  The incidence of necrotizing enterocolitis
Spontaneous intestinal perforation | Duration of hospitalization, an average of 8-15 weeks
  The incidence of spontaneous intestinal perforation
Bronchopulmonary dysplasia | At timepoint of reached 36 gestational weeks of the neonate
  Incidence of bronchopulmonary dysplasia
Intraventricular and periventricular haemorrhage | Duration of hospitalization, an average of 8-15 weeks
  The incidence of intraventricular and periventricular haemorrhage (stage I-IV)
Retinopathy of prematurity | Duration of hospitalization, an average of 8-15 weeks
  Incidence of retinopathy of prematurity (stage I-V)
Neurodevelopment | Follow up at 24 months of corrected age of the child
  Assessment of neurodevelopmental outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zbynek Stranak, MD, Study Chair — Institute for the Care of Mother and Child in Prague
Locations (2):
- Institute for the Care of Mother and Child, Prague, Czechia
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Available on request after publication of study results

REFERENCES:
- [Derived] Branagan A, Murphy C, O'Sullivan A, Bodnarova I, Feyereislova S, Berka I, Miletin J, Stranak Z. Influence of gastric residual assessment in preterm neonates on time to achieve enteral feeding (the GRASS trial)-Multi-centre, assessor-blinded randomised clinical trial. Eur J Pediatr. 2024 May;183(5):2325-2332. doi: 10.1007/s00431-024-05483-w. Epub 2024 Mar 1. PMID 38427039